CLINICAL TRIAL: NCT03808701
Title: Recombinant Anti-EGFR Monoclonal Antibody（SCT200） in Patients With Advanced Squamous Non-small Cell Lung Cancer : a Phase Ib, Open-label, Multicenter Study
Brief Title: Efficacy and Safety of SCT200 in Patients With Advanced Squamous Non-small Cell Lung Cancer
Acronym: sNSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT200-D101
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Advanced Squamous Non-small Cell Lung Cancer
Keywords: SCT200; Squamous non-small cell Lung cancer; NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose group (Experimental): Initially, 9.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 12.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Interventions: Drug: SCT200
- HIGH dose group (Experimental): Initially,12.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 15.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Interventions: Drug: SCT200

INTERVENTIONS:
Drug: SCT200 — Recombinant Anti-EGFR Monoclonal Antibody

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-EGFR monoclonal antibody（SCT200）in patients with advanced squamous non-small cell lung cancer treated after failure of Two chemotherapy regimens (including Platinum-based drugs).

DETAILED DESCRIPTION:
This open label multicenter phase Ib study is designed to evaluate Objective Response Rate (ORR) in Squamous non-small cell Lung cancer treated with anti-EGFR monoclonal antibody SCT200.

ELIGIBILITY:
Inclusion Criteria:

Able to provide written informed consent and can understand and comply with the requirements of the study;

Men/Women from 18 to 75 years old;

Life expectancy of longer than 3 months ( clinical assessment);

With an Eastern Cooperative Oncology Group (ECOG) performance status 0-1;

Histological or cytological diagnosis of Squamous non-small cell Lung cancer;

Locally advanced or metastatic NSCLC(stage IIIB/IV or recurrent NSCLC that do not meet the criteria for radical radiotherapy and chemotherapy，Tumor stage will be classified according to UICC/AJCC staging system version 8).Participants has received at least two previous chemotherapy regimens for treatment failure (including disease progression and unacceptable toxic and side effects).

Note: a. first-line chemotherapy must be a platinum-containing two-drug regimen;b. Prior adjuvant/neoadjuvant chemotherapy is permitted.If recurrence or metastasis occurs during or within 6 months after the completion of adjuvant/neoadjuvant chemotherapy, it is considered that adjuvant/neoadjuvant chemotherapy is a first-line systemic chemotherapy failure for advanced disease." According to RECIST 1.1 , patients must have at least one measurable lesion that can be accurately assessed at baseline.

Adequate organ and marrow function as defined below:

Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 75×109/L; Hemoglobin greater than/equal to 80g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 3 times ULN, or less than/equal to 5 times ULN if known liver metastases; Total bilirubin less than/equal to 1.5 within institutional limit of normal (ULN); Serum creatinine less than/equal to 1.5 times ULN; Electrolyte: magnesium greater than/equal to normal.

-

Exclusion Criteria:

Patients are allergic to antibodies or other components contained in the test drugs;

Symptomatic metastatic central nervous system and/or cancerous meningitis.(After treatment for brain metastasis, disease should be stable and last for at least 4 weeks prior to the first study administration, not requiring for steroid or anticonvulsant therapy,Subjects with stable neurological symptoms may be enrolled ).For stable asymptomatic brain metastases that have been treated with radiotherapy, at least one other site besides the brain metastasis can be measured ,The subject can be enrolled, but the interval between the last radiotherapy should be more than 4 weeks..

Subject receiving bisphosphonate or denosumab treatment for bone metastases was initiated within 28 days prior to study. (If the subject has received bisphosphonate or denosumab treatment prior to study and showing stable time less than 28 days,the subject is allowed to use it.) If the ongoing bisphosphonate therapy dose is considered to be increased or bisphosphonate therapy is initiated due to the aggravation of bone pain, researchers should confirm whether the subject has PD according to the RECIST1.1 version.

Patients with other primary malignancies, except for before 5 years or more, malignant lesions had been treated with therapeutic measures and no known active lesions existed, and the researchers judged that the risk of recurrence was low;Non-melanoma skin cancer treated adequately without evidence of disease progression; cervical carcinoma in situ after adequate treatment;Prostate intraepithelial neoplasm, no evidence of recurrence of prostate cancer;

Patients administrated EGFR target treatment including EGFR TKI agent or anti- EGFR monoclonal antibody;

Within 4 weeks, patients received anti-tumor drugs (such as chemotherapy, hormone therapy, immune therapy, the antibody therapy, radiotherapy) or research drugs(42 days for nitrosourea or mitomycin C), or patients with grade 2 or more adverse reaction caused by previous anti-tumor therapy(except alopecia or neurotoxicity grade 2 or less);

Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices.

"Patients received major surgery(such as general anesthesia ) within 4 weeks ,or subjects did not recovered from the injury associated with the surgery.

Note: surgery requiring local/epidural anesthesia must have been completed for at least 72 hours and subjects must have recovered before starting the study medication.Skin biopsy under local anesthesia has been completed for at least 1 hour."

Patients treated with EPO, G-CSF or GM-CSF before enrollment 2 weeks.

Patients who have clinically significant cardiovascular disease (defined as unstable angina pectoris, symptomatic congestive heart failure (NYHA, greater than II), uncontrollable severe arrhythmia); Patients occurred myocardial infarction within 6 months.

Patients who have interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or on baseline chest CT or MRI reminder ILD .

Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);

Patients with active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, HBV DNA ≥104 or ≥ 2000IU/ml, HCV RNA≥15IU/ml); HIV antibody positive (if there is no clinical evidence suggesting that there may be HIV infection, there is no need to detect);

Patients with uncontrolled active infections before enrollment 2 weeks (except simple urinary tract infection or upper respiratory tract infection);

Pregnant or lactating women(Serum test must be negative within 7 days prior to study enrollment)

Patients((including male or female subjects) who were not willing to accept effective contraceptive measures( intrauterine device, prophylactic or condom)during treatment and within 6 months after treatment;

Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator，such as inability to comply with study and/or follow-up procedures;

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.

SECONDARY OUTCOMES:
Progress Free Survival ( PFS) | 1 year
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 criteria.
Disease control rate (DCR) | 1 year
  The achievement of any a stable response（SD）, partial response (PR) or complete response (CR), according to RECIST v1.1 criteria.
Duration of response (DOR) | 1 year
  DOR is defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1, until the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Overall survival (OS) | 1 year
  OS is defined as time from first dose of SCT200 until the date of death from any cause.
AE | 1 year
  AE are assessed according to NCI CTCAE v4.03.
Evaluation of immunogenicity | 1 year
  Serum SCT200 antibody levels were measured before and after administration.
exploratory analysis | 1 year
  To explore the possible correlation between EGFR and/or related gene expression and disease prognosis and therapeutic efficacy

CONTACTS AND LOCATIONS:
Overall Officials: CHENG YING, MD, Principal Investigator — Jilin Provincial Cancer Hospital